CLINICAL TRIAL: NCT04456660
Title: Markers of Ultrasound, Immunologic & Serum Factors in the Comprehensive Analysis of Risks for Early Pregnancy Loss.
Brief Title: Comprehensive Assessment of Risks for Miscarriage.
Acronym: MIS-CARE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Orthogyn Medical Center, Bulgaria (Other)
Responsible Party: Principal Investigator, Petar Ignatov, Assist. Prof. Petar Ignatov, MD, Ph.D., Orthogyn Medical Center, Bulgaria
Other Study IDs: MIS-CARE
Record Dates: First submitted 2020-06-25; First posted 2020-07-02 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Spontaneous Abortion
MeSH Terms: conditions — Abortion, Spontaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control group: Monitoring of pregnancy, including data on:
  * maternal age and other demographic characteristics;
  * ultrasound measurement of fetal heart rate (FHR) and crown-rump length (CRL)
- sFlt-1, Doppler and NK cells types group: Monitoring of pregnancy, including data on:
  * maternal age and other demographic characteristics;
  * ultrasound measurement of fetal heart rate (FHR) and crown-rump length (CRL), uterine arteries PI, and other parameters;
  * measurement of serum sFlt-1, PLGF, and glycodelin-A levels, as well as other parameters;
  * measurement of CD16+, CD56+, and other subpopulations of NK cells;
  Interventions: Diagnostic Test: Markers of ultrasound; Diagnostic Test: Immunologic factors; Diagnostic Test: Serum factors

INTERVENTIONS:
Diagnostic Test: Markers of ultrasound — CRL, HR, and other ultrasound measurements.
  Groups: sFlt-1, Doppler and NK cells types group
Diagnostic Test: Immunologic factors — Measurement of NK cells subpopulations types in the maternal serum
  Groups: sFlt-1, Doppler and NK cells types group
Diagnostic Test: Serum factors — Measuring the maternal serum concentration of sFlt-1, PLGF, glycodelin-A, and other substances.
  Groups: sFlt-1, Doppler and NK cells types group

SUMMARY:
This study aims to determine the role of serum biomarkers and placental bloodflow in the comprehensive evaluation of the risk for spontaneous abortion

DETAILED DESCRIPTION:
To study the added value (if any) of combining serum markers, immunologic factors, and ultrasound parameters in comprehensively evaluating the risk for spontaneous abortion.

ELIGIBILITY:
Inclusion Criteria:

* visualized fetal structures in utero & heart pulsations until 8th week of gestation
* normal THS/T4 levels
* no uterine malformations
* BMI < 27
* signed informed consent

Exclusion Criteria:

* fetal structures in utero & heart pulsations not visualized until the 8th week of gestation
* elevated THS/T4 levels
* uterine malformations
* BMI > 27

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Pregnant women between 18 and 50 years of age.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-06-20 (Actual); Primary Completion 2023-11-20 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Occurence of a spontaneous abortion | Up to 24 weeks of gestation
  Absent heart rate pulsations on an ultrasound scan

CONTACTS AND LOCATIONS:
Overall Officials: Petar N Ignatov, PhD, Principal Investigator — Orthogyn Medical Center
Locations (1):
- Orthogyn Medical and Dental Center, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: No